CLINICAL TRIAL: NCT05041764
Title: A Comparison Between Individual and Wastewater SARS-CoV2 RNA Sequencing
Brief Title: RNA Sequencing of Individual Versus Wastewater - SARS-CoV2
Acronym: Cagablea
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: 21DSP-IPMC01
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCR positive: samples that are positive for the detection of SARS-CoV2. The SARS-CoV2 sequence of positive samples is provided, together with an indication about patient's neigborhood, corresponding to one of the 21 different spots which wastewater was analyzed
  Interventions: Other: NO INTERVENTION
- PCR negative: samples that are p negative for the detection of SARS-CoV2. T
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — No INTERVENTION

SUMMARY:
The aim is to compare the percentage of the different SARS-CoV2 lineages that are detected in wastewater samples with matched clinical samples. About 1,400 swab samples from patients living in Nice were tested by Biogroup between Oct 19th and Oct 23rd (Week 43 of 2020). The sequence of 81 PCR positive samples, corresponding to all samples that were unambiguously assigned to one of the wastewater catchment areas and their lineage was determined. These values were compared to values measured in wastewater.

ELIGIBILITY:
Inclusion Criteria:

* whole population tested in Nice during W43 of 2020

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nice population
Sampling Method: Probability Sample
Enrollment: 1409 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
RTqPCR result | 1 month
  positive ou negative result to SAR-Cov2
SARS-CoV2 sequence | 1 month
  analyse of SARS-CoV2 sequence (in the case of positive samples)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nice Hospital, Nice
  - Ipmc . Cnrs, Sophia Antipolis

IPD SHARING:
Plan to Share IPD: Undecided